CLINICAL TRIAL: NCT03914768
Title: Immune Modulatory DC Vaccine Against Diffuse Intrinsic Pontine Glioma (DIPG) and Glioblastoma (GBM)
Brief Title: Immune Modulatory DC Vaccine Against Brain Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-19001
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Diffuse Intrinsic Pontine Glioma or Glioblastoma
Keywords: DC vaccine therapy; DIPG; GBM; neoantigen
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioblastoma

STUDY DESIGN:
Intervention Model Description: Patients with DIPG or GBM will be treated with immunomodulatory DC vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunomodulatory DC vaccine to target DIPG and GBM (Experimental): Patients will receive immune modulatory treatment consisting of cyclophosphamide (200 mg/m2) and bevacizumab (15 mg/kg), before and after DC vaccine injection, respectively.
  Interventions: Biological: Immunomodulatory DC vaccine to target DIPG and GBM

INTERVENTIONS:
Biological: Immunomodulatory DC vaccine to target DIPG and GBM — This study will inject DC vaccine cells near lymphoid tissue close to the tumor. The patient will receive intravenous cyclophosphamide (200 mg/m2) or oral (cytoxan) before the vaccine, followed by DC vaccine and intravenous bevacizumab (15 mg/kg) the next day. The cells will be repeatedly infused every month for six consecutive months depending on the response and the condition of the patient. The amount of DC vaccine cells per injection is based on prior report at 5-10x106. An initial dose escalation scheme will be imposed.

SUMMARY:
This study is designed to treat patients who have been diagnosed with brain cancer, including glioblastoma (GBM) and diffuse intrinsic pontine glioma (DIPG). The treatment uses immunomodulatory vaccine generated by autologous dendritic cells (DCs) pulsed with genetically modified tumor cells or tumor-related antigens including neoantigens to inject into patients. Vaccine-induced T cell responses have been associated with improved survival. The study will evaluate the safety and potential benefit of the novel immunomodulatory DC vaccines.

DETAILED DESCRIPTION:
Diffuse intrinsic pontine glioma (DIPG) or glioblastoma (GBM) is an aggressive malignancy. DIPG mainly occurs in the ventral pontine of childhood. The overall median survival time is 9 to 11 months. The 2-year survival rate is less than 10%. Thus DIPG has become one of the most fatal diseases in children. These tumors invade and infiltrate the surrounding brain, making complete surgical excision impossible. Several studies focused on the identification of GBM or DIPG-specific antigens and evaluated their potential for vaccine application. Immunomodulatory DC vaccines based on ex vivo genetic modifications in combination with known tumor-specific antigens may substantially enhance the activation potential of tumor-specific T cells with improved benefit to patients.

Although certain antigens are highly specific in DIPG or GBM, existing immune tolerance suppresses anti-tumor immunity in cancer patients. To induce anti-cancer immune response in patients, ex vivo modification of immune modulatory antigens or immune cells will be necessary. Advanced whole exome sequencing has been developed to identify specific mutations in tumors and predict best-fit MHC-specific neoepitopes for T cell activation. In this study we will investigate novel DC vaccines based on autologous DCs pulsed with genetically modified tumor cells or related antigens such as neoantigens to induce a strong anti-tumor immunity. Early studies of DC-based vaccines targeting gliomas have shown acceptable safety and low toxicity profile. This is a multi-center randomized Phase I study to evaluate safety of novel DC vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Abilities to understand and the willingness to provide written informed consent. Assent will be obtained when appropriate based on the subjects age;
2. Patients are ≥ 6 months and ≤ 80 years old;
3. DIPG or GBM patients with existing or measurable tumors in the brain. Patients have received standard care of medication, such as gross total resection with concurrent radio chemotherapy (~54 - 60 Gy, TMZ);
4. Patients with adequate neurological function and epileptic symptoms that are well controlled;
5. Observing the condition after surgery or without surgery;
6. Karnofsky performance score (KPS) ≥ 60;Life expectancy >3 months;
7. Important organ function is satisfied: Cardiac ultrasound indicates a cardiac ejection fraction ≥50%; and there is no obvious abnormality in the electrocardiogram; blood oxygen saturation ≥90%; creatinine <2.5 times normal range; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 times normal range; Total bilirubin ≤ 2.0 mg / dl; Hgb (hemoglobin) ≥ 80g / L;
8. Peripheral blood absolute lymphocyte count must be above 0.8×10^9/L;
9. Adequate Neurologic Function Defined as: Patients with seizure disorder may be enrolled if seizure disorder is well controlled;
10. Patients must be willing to follow the orders of doctors.

Exclusion Criteria:

1. A prior history of gliadel implantation 4 weeks before this study start or antibody based therapies;
2. The patient was still using dexamethasone at a dose greater than 4 mg/day during mononuclear cell collection;
3. Patients have a history of autoimmune diseases or other diseases requiring long-term use of hormones or immunosuppressive drugs;
4. Patients with a history of allergies or allergies to immune cells and adjuvants of cellular products;
5. Active infection with fever;
6. Patients with neutropenia (> 10 days) that are difficult to correct after treatment;
7. Infection with bacteria, fungi or viruses, uncontrolled;
8. Patients with HIV and those living with active HBV and HCV;
9. Pregnant, pregnant and lactating women;
10. Important organ failure (heart, liver, kidney, lung);
11. Patients who had previously been treated with cell therapy but were ineffective after physical examination were discussed and confirmed by team experts and were not suitable for re-treatment;
12. Anything that researchers believe may increase the risk of subjects or interfere with test results.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion of autologous immunomodulatory DC Vaccine is assessed by the NCI CTCAE V4.0 criteria. | 2 years
  Safety of the vaccine will be assessed by monitoring for adverse events (AEs) based on scheduled laboratory assessments.
Overall survival (OS) at 12 months (OS12). | 12 months
  OS12 will be the clinical efficacy primary endpoint. For subjects who are still alive at 12 months, OS12 will be censored at the last contact date. OS will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Treatment response rate of DIPG or GBM | 6 months]
  Defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) based on brain MRI imaging analysis.
Overall survival Rate | 1 year follow up
  Percentage of participants with objective response as determined by the investigator based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Progression-free survival rate | 1 years
  Progression-free Survival (PFS) as determined by the investigator based on RECIST v1.1
ELISPOT or antigen specific functional assays for evaluation of antigen specific immune response in patients | 1 year
  Tumor antigen specific immune response in the peripheral blood evaluated by ELISPOT or antigen specific functional assays.
Magnetic resonance imaging for evaluation of disease progression and prognosis | 1 years
  The prognosis of GBM or DIPG will be determined by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (3):
- China (3):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Department of Neurosurgery, Shenzhen Hospital, Southern Medical University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No